CLINICAL TRIAL: NCT03731221
Title: A Comparison of Combined Pectoral Fascial Plane and Serratus Anterior Plane Blocks With Bupivacaine HCL With and Without Liposomal Bupivacaine for Video Assisted Thoracic Surgery
Brief Title: Pectoral Fascial Plane and Serratus Anterior Plane Blocks With Bupivacaine v. Liposomal Bupivacaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Donn Marciniak, Enterprise Chair, Dept of Intensive Care and Resuscitation, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-981
Record Dates: First submitted 2018-10-22; First posted 2018-11-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Video Assisted Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: Patients will be randomized the day of surgery upon presentation to the operating room to either a treatment group (PECSII/SAP blocks with bupivacaine HCl plus liposomal bupivacaine) or a control group (PECSII/SAP blocks with bupivacaine HCl plus preservative free normal saline) using secure web-based randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthesiologists will not be blinded to the intervention, but all outcomes will be assessed by research personnel who are blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupi HCl plus liposomal bupi (Experimental): PECSII/SAP blocks with bupivacaine HCl plus liposomal bupivacaine
  Interventions: Drug: Bupi HCI and lipo bupi
- Bupi HCl plus saline (Active Comparator): PECSII/SAP blocks with bupivacaine HCl plus preservative free normal saline
  Interventions: Drug: Bupi HCI

INTERVENTIONS:
Drug: Bupi HCI and lipo bupi — The local anesthetic (LA) used for the PECS II or serratus plane blocks will be a 0.5% bupivacaine HCL, not to exceed 2.5mg/kg or up to 150mg. The LA solution can be diluted with preservative free normal saline for smaller patients to allow for appropriate volume of injection. Treatment patients will also be given liposomal bupivacaine (EXPAREL, Pacira Pharmaceuticals, Inc. San Diego, CA) in a dose of 266 mg in 20 ml can be safely combined with bupivacaine HCL at a ratio not exceeding 2:1, but cannot be combined with other local anesthetics due to the concern of rapid release of encapsulated bupivacaine and subsequent local anesthetic toxicity.
  Other Names: Bupi and lipo bupi
  Arms: Bupi HCl plus liposomal bupi
Drug: Bupi HCI — The LA used for the blocks will be a 0.5% bupivacaine HCL, not to exceed 2.5mg/kg or up to 150mg. The LA solution can be diluted with preservative free normal saline for smaller patients to allow for appropriate volume of injection. Control patients will have preservative free normal saline mixed with 0.5% bupivacaine HCL and all patients will have a total block solution volume of 60 ml.
  Other Names: Control
  Arms: Bupi HCl plus saline

SUMMARY:
Patients will be randomized the day of surgery upon presentation to the operating room to either a treatment group (PECSII/SAP blocks with bupivacaine HCl plus liposomal bupivacaine) or a control group (PECSII/SAP blocks with bupivacaine HCl plus preservative free normal saline) using secure web-based randomization. Assignments will be based on computer-generated code. Clinicians will not be blinded to the intervention, but all outcomes will be assessed by research personnel who are blinded to the group assignment.

DETAILED DESCRIPTION:
Anesthetic care will be performed in a usual manner in Cleveland Clinic thoracic surgical patients. This includes the use of standard ASA monitors and may include the use of arterial or central venous pressure monitoring, trans-esophageal echocardiography, and lung isolation using a bronchial blocker or a double lumen endotracheal tube. Medication administration for induction and maintenance of anesthesia will also be consistent with usual care and will include intravenous opioids such as fentanyl and hydromorphone. Intravenous lidocaine boluses will not be administered upon induction of anesthesia. Pressure control ventilation will be utilized with a tidal volume not exceeding 6-10 ml/kg ideal body weight during two-lung ventilation and 5-7 ml/kg ideal body weight during one-lung ventilation. A conservative fluid management strategy will be employed in all cases. Patients not extubated at the end of the procedure will be sedated with propofol. Surgical procedures will be performed in their usual manner.

The anatomic basis for chest wall analgesia has been described in detail previously. The investigators describe the conduct of the blocks as used for VATS procedures at the investigator's institution. The patients randomized to the treatment group will all receive PECSII and serratus blocks containing bupivacaine HCl and liposomal bupivacaine. The control group will receive PECSII and serratus blocks with bupivacaine HCl adjusted to a similar volume. The PECS/serratus blocks will be performed with the patient under the general anesthesia and before incision. If this is not possible due to surgical urgency, the block will be placed at end of surgery.

Patients will be positioned supine, and prepped and draped in a sterile fashion. An ultrasound probe will be placed just below the clavicle in the mid-clavicular line.

For the PECS II block, the probe will be scanned inferiorly and laterally until the plane between the pectoralis minor and serratus muscle is identified. The serratus muscle can be clearly seen coursing over the ribs, while the intercostal muscles are seen in the interspaces between the ribs. Once the plane is identified the needle is again advanced in an "in-plane" fashion. Once the needle location is confirmed by normal saline hydro-dissection, a 15-20 cc of local anesthetic solution is administered into the space.

With the patient in a supine position, a back roll will be placed under the operative side to achieve a slightly lateral tilt. The arm is abducted to expose the costal margin. The positioning and prepping is done prior to the PECS block to avoid repositioning. The ultrasound probe is scanned laterally from the pectoralis to the axillary region at approximately the level of the 5th rib. The plane between the serratus muscle and the latissimus dorsi muscle is identified and the needle advanced in an "in-plane" fashion until the tip is between the muscles (superficial SAP block). A small bolus of 0.5 cc of normal saline is used for hydro-dissection of the tissue planes to confirm that the needle is not intramuscular. The needle is then aspirated every 5 cc as 40 cc of local anesthetic solution is deposited into the plane. As these are field blocks, adequate volume of infiltration is important in achieving optimal analgesia.

The LA used for the blocks will be a 0.5% bupivacaine HCL, not to exceed 2.5mg/kg or up to 150mg. The LA solution can be diluted with preservative free normal saline for smaller patients to allow for appropriate volume of injection. Typically the block has duration of action of less than 12 hours after infiltration.34 Treatment patients will also be given liposomal bupivacaine (EXPAREL, Pacira Pharmaceuticals, Inc. San Diego, CA) in a dose of 266 mg in 20 ml can be safely combined with bupivacaine HCL at a ratio not exceeding 2:1, but cannot be combined with other local anesthetics due to the concern of rapid release of encapsulated bupivacaine and subsequent local anesthetic toxicity.35 Control patients will have preservative free normal saline mixed with 0.5% bupivacaine HCL and all patients will have a total block solution volume of 60 ml.

Liposomal bupivacaine dosing is not weight based and the full 266-mg bottle can be administered to adult thoracic patients. A maximum of 150mg bupivacaine HCl can be mixed with Exparel. This equates to one 30-mL bottle of 0.5% bupivacaine HCl or two (2) bottles of 0.25% bupivacaine HCl. If a higher volume of the LA is needed a 10 ml of normal saline can be added to the mixture of bupivacaine HCL and liposomal bupivacaine. Thus patients ≥60 kg will receive 150 mg of bupivacaine HCL, while patients weighing <60 kg need to have the bupivacaine dose calculated but can still receive full 20 ml of Exparel.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-85 years of age
2. Procedures using thoracic access ports or miniature thoracotomy incisions such as video assisted thoracic surgical (VATS) or robotic anatomic pulmonary resection (lobectomy, bilobectomy, and segmentectomy)

Exclusion Criteria:

1. Weight less than 50 kg
2. Pregnancy or lactation
3. Emergency surgery and patients transferred from the ICU to the operating room
4. Redo thoracic surgery or post-operative reoperation within 72 hours of index procedure (including minor chest wall procedures including tube thoracostomy, thoracentesis or percutaneous drain placement)
5. Anticipated endotracheal intubation > 24 hours
6. Non-study nerve block that provides analgesia to the intercostal nerves
7. Active systemic or cardiopulmonary infection
8. Mechanical circulatory support devices
9. Allergy or contraindication to study local anesthetics
10. More than 15 mg/day morphine equivalents on at least 15 of the 30 preoperative days
11. Poorly controlled psychiatric disorders
12. Clinically important current neurologic deficit e.g. spinal cord injury, paralysis of extremity, any neurologic deficit in the region of the block
13. Active liver disease or cirrhosis
14. Pacemaker generator or breast implants ipsilateral to surgery
15. Previous participation in this study
16. eGFR <30 or chronic kidney disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Overall benefit of analgesia score | Postoperative day 3
  The overall benefit of analgesia score (OBAS) is based on 7 questions and ranges from 0 to 28 points

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on a collaborative basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of main paper.
Access Criteria: IPD will be shared on a collaborative basis.